CLINICAL TRIAL: NCT03638661
Title: Effect of Immune-enhancing Enteral Nutrition Formula Enriched With Vegetable Derived n-3 Fatty Acids on NK Cell Activity in Hospitalized Patients for Rehabilitation
Brief Title: n-3 Fatty Acids in Enteral Formula on NK Cell Activity
Acronym: YS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, Principal Investigator, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YS
Record Dates: First submitted 2018-08-06; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Enteral Nutrition
MeSH Terms: interventions — Vegetables; Linseed Oil; Soybean Oil

STUDY DESIGN:
Who Masked: Participant
Masking Description: The ready-to-use soybean used formula and n3EN formula had identical packaging with no differences in appearance, texture, or smell.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- n-3 fatty acid enriched formula (Experimental): Those assigned to the n3EN group received vegetable n-3 fatty acid enriched formula by tube feeding (product; Yonsei Dairy Co., Seoul, South Korea).
  vegetable (canola, flaxseed) derived n-3 fatty acid
  Interventions: Dietary Supplement: vegetable (canola, flaxseed) derived n-3 fatty acid
- soybean oil used formula (Placebo Comparator): Patients assigned to the control group received a soybean used formula by tube feeding.
  soybean used formula
  Interventions: Dietary Supplement: soybean oil

INTERVENTIONS:
Dietary Supplement: vegetable (canola, flaxseed) derived n-3 fatty acid — vegetable (canola, flaxseed) derived n-3 fatty acid was used for fat source.
  Arms: n-3 fatty acid enriched formula
Dietary Supplement: soybean oil — soybean oil used formula
  Arms: soybean oil used formula

SUMMARY:
The aim of our study was to investigate the NK cell activity alternations and related cytokine changes in comparison with soybean oil used formula (control) and the canola and flaxseed oil used n-3 fatty acid enriched formula (n3EN, test) with non-surgical hospitalized patients for rehabilitation.

DETAILED DESCRIPTION:
Patients were randomized to receive one of two types of enteral nutrition formula: soybean oil used enteral nutrition (control), vegetable (canola, flaxseed) derived n-3 fatty acid enriched enteral nutrition (n3EN). Blood samples were collected on the first day and 14 days after consumption of each formula and anthropometric parameters were collected. Hematology and biochemical values were analyzed and NK cell activities and serum cytokine productions were measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were admitted to the Severance Hospital Rehabilitation Department , enteral tube feeding patient, Adult male and female patients aged 19 years and over, Patients who signed the consent form

Exclusion Criteria:

* Patient with nausea
* Patients with hepatic impairment (total bilirubin concentration> 3.5 mg / dl)
* Patients with renal impairment (serum creatinine concentration> 3 mg / dl or requiring peritoneal or hemodialysis) diabetic patients
* Patients who are undergoing chemotherapy or who are within 1 month of the end of chemotherapy
* Patients whose life expectancy is less than 1 month
* Pregnant women and women who are pregnant

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
NK cell activity | Baseline
  NK cell activity (%)

SECONDARY OUTCOMES:
cytokine values | Baseline
  (IL-12, IFN-γ, IL-1β , IL-6 and TNF-α)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT03638661/Prot_SAP_000.pdf